CLINICAL TRIAL: NCT02293629
Title: A Randomized, Double-Blinded, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Pharmacokinetics, and Target Engagement of BMS-986147 in Healthy Subjects
Brief Title: A Single and Multiple Ascending Dose Study to Evaluate the Safety, Pharmacokinetics, and Target Engagement of BMS-986147 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: IM008-003
Record Dates: First submitted 2014-11-14; First posted 2014-11-18 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- A1: BMS-986147 or Placebo matching BMS-986147 (Placebo Comparator): Single oral dose as specified
  Interventions: Drug: BMS-986147; Drug: Placebo matching BMS-986147
- A2: BMS-986147 or Placebo matching BMS-986147 (Placebo Comparator): Single oral dose as specified
  Interventions: Drug: BMS-986147; Drug: Placebo matching BMS-986147
- A3: BMS-986147 or Placebo matching BMS-986147 (Placebo Comparator): Single oral dose as specified
  Interventions: Drug: BMS-986147; Drug: Placebo matching BMS-986147
- B1: BMS-986147 or Placebo matching BMS-986147 (Active Comparator): Daily oral dose as specified
  Interventions: Drug: BMS-986147; Drug: Placebo matching BMS-986147
- B2: BMS-986147 or Placebo matching BMS-986147 (Active Comparator): Daily oral dose as specified
  Interventions: Drug: BMS-986147; Drug: Placebo matching BMS-986147

INTERVENTIONS:
Drug: BMS-986147
Drug: Placebo matching BMS-986147

SUMMARY:
This is the first clinical study with the BMS-986147 compound in healthy subjects. The purpose of this study is to guide the dose range and dose frequency for future studies with BMS-986147 and will provide guidelines for selection of a potentially effective dose in patients.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy men and women, ages 18 to 45 years
* Subjects must not have clinically significant deviation from normal: medical history, physical examination, ECGs and laboratory evaluations
* Women of child bearing potential are eligible for enrollment.
* Women must have a negative pregnancy test

Exclusion Criteria:

* Evidence of organ dysfunction
* Any significant acute or chronic medical illness
* Inability to: tolerate oral medications, be venipunctured

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single oral dose of BMS-986147 based on incidence of AEs, serious AEs, AEs leading to discontinuation, and death as well as marked abnormalities in clinical laboratory tests, vital sign measurements, and physical examinations | Up to 30 days post last dose of study drug
  Adverse event (AE)
Safety and tolerability of multiple oral dose of BMS-986147 based on incidence of AEs, serious AEs, AEs leading to discontinuation, and death as well as marked abnormalities in clinical laboratory tests, vital sign measurements, and physical examinations | Up to 30 days post last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Wcct Global, Llc, Cypress, California, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx